CLINICAL TRIAL: NCT01495624
Title: The Effect of Systemic or Perineural Dexamethasone on the Duration of Interscalene Nerve Blocks With Ropivacaine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual insufficient to complete study in a feasible time frame
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kenneth Cummings III, MD, MS, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-1048
Record Dates: First submitted 2011-12-12; First posted 2011-12-20 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Duration of Interscalene Block
Keywords: rotator cuff repair; capsular shift; shoulder arthroplasty; subacromial decompression; 18 and 75 years
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine with perineural dexamethasone (Placebo Comparator): 30 ml 0.5% ropivacaine plus dexamethasone 8 mg (2 ml) mixed with the local anesthetic with 2 ml normal saline given intravenously (systemic placebo);
  Interventions: Other: ropivacaine plus dexamethasone anesthetic
- Ropivacaine with systemic steroid (Active Comparator): 30 ml 0.5% ropivacaine for interscalene block mixed with 2 ml normal saline (perineural placebo) plus dexamethasone 8 mg (2 ml) administered systemically.
  Interventions: Other: ropivacaine plus saline plus dexamethasone anesthetic

INTERVENTIONS:
Other: ropivacaine plus dexamethasone anesthetic — Subjects will receive interscalen block comprised of 30 ml 0.5% ropivacaine plus dexamethasone 8 mg (2 ml) mixed with the local anesthetic with 2 ml normal saline given intravenously (systemic placebo);
  Arms: Ropivacaine with perineural dexamethasone
Other: ropivacaine plus saline plus dexamethasone anesthetic — Subjects will receive interscalen block with 30 ml 0.5% ropivacaine for interscalene block mixed with 2 ml normal saline (perineural placebo) plus dexamethasone 8 mg (2 ml) administered systemically.
  Arms: Ropivacaine with systemic steroid

SUMMARY:
Patients undergoing rotator cuff repair or subacromial decompression at the investigators institution are frequently hospitalized overnight due to inadequate pain relief after resolution of interscalene brachial plexus blocks. For ropivacaine 0.5%, the investigators usual local anesthetic, previous studies report an analgesic duration of 11.1 ± 5 hours without epinephrine and approximately 12 hours with epinephrine. Consequently, a method of prolonging analgesia from a brachial plexus block without the extra equipment and logistical difficulties of indwelling catheters would benefit both patients and caregivers. A potential approach is use of adjuvant drugs that prolong block duration when added to the local anesthetic.

In addition to the usual adjuvant anesthetic drugs, investigators have begun to evaluate glucocorticoids as adjuvants for regional anesthesia. Known for their anti-inflammatory, analgesic, immunosuppressive, and antiemetic properties, these corticosteroids exert their effects by inhibition of phospholipase A2 as well as changes in cell function induced by glucocorticoid receptor activation. Although associated with significant toxicity when administered in large doses for long periods, emerging literature suggests that a single perioperative dose of glucocorticoid is safe. Several studies, including a recent trial at the investigators institution, have demonstrated the efficacy of dexamethasone in prolonging regional anesthetics. Available data thus suggest that combining glucocorticoids with local anesthetics prolongs block duration. However, systemic glucocorticoids have also been shown to reduce postoperative pain. This raises the question whether the beneficial effects of adding glucocorticoid to a regional anesthetic is solely due to local effect or is mediated at least in part by systemic action. Previous trials, however, have not addressed this important issue. If this beneficial effect of analgesic duration is mediated by systemic action, adding dexamethasone to the local anesthetic mixture may be unnecessary. Although no study has reported neurotoxicity from perineural dexamethasone and laboratory data appear to confirm the safety of this route, achieving similar results with more conventional administration would be desirable for two reasons. First, conventional intravenous dosing is convenient, useful for other reasons (for example, postoperative nausea prophylaxis), and well-studied. Second, equivalent (or not equivalent) results from systemic dosing would provide valuable information about the mechanism behind dexamethasone's effect on block duration.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing shoulder procedures such as

* Rotator cuff repair
* Capsular shift
* Shoulder arthroplasty
* Subacromial decompression

  • Exclusion Criteria:
  * Contraindications to interscalene block
* Coagulopathy
* Infection at the needle insertion site
* Moderate to severe chronic obstructive pulmonary disease (COPD)
* Contralateral pneumothorax or diaphragmatic paralysis

  * Pregnancy
  * Preexisting neuropathy involving the surgical limb
  * Systemic glucocorticoid treatment (for at least one week) within six months of surgery
  * Routine opioid use (greater than 30 mg oxycodone per day or equivalent)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
duration of interscalene nerve block | Day one
  The clinical duration of the interscalene nerve block, which will be measured by time from onset of sensory block until first administration of analgesic medication or requirement for initiation of the perineural catheter infusion.

SECONDARY OUTCOMES:
increase in shoulder discomfort | as reported in minutes after procedure, day one
  time to a noticeable increase in shoulder discomfort, maximum VRS with rest and movement, and total opioid consumption.
maximum VRS (Verbal Response Score) with rest | upon admission to PACU through post operative day 2, post operative day 14
  time to a noticeable increase in shoulder discomfort, maximum VRS (Verbal Response Score) with rest and movement, and total opioid consumption.
Verbal Response Score (VRS) with movement | upon admission daily through post operative day 2, post operative day 14
  time to a noticeable increase in shoulder discomfort, maximum VRS with rest and movement, and total opioid consumption.
total opioid consumption | daily through post operative day 2
  time to a noticeable increase in shoulder discomfort, maximum VRS with rest and movement, and total opioid consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cummings, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Bei T, Liu J, Huang Q, Wu J, Zhao J. Perineural Versus Intravenous Dexamethasone for Brachial Plexus Block: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Pain Physician. 2021 Sep;24(6):E693-E707. PMID 34554686